CLINICAL TRIAL: NCT01321879
Title: Phase II, Open-Label Pilot Study to Evaluate the Safety and Efficacy of Telavancin in the Treatment of Gram Positive Bloodstream Infections in Cancer Patients
Brief Title: Study to Evaluate the Safety and Efficacy of Telavancin in the Treatment of Gram Positive Bloodstream Infections in Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0454; NCI-2011-00752 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2011-03-17; First posted 2011-03-24 (Estimated); Results first posted 2019-12-27 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Infection; Bacteremia
Keywords: Gram Positive Bloodstream Infections; Sepsis; Staphylococcus aureus; Enterococci; Streptococci; Pneumococci; Corynebacterium; Propionibacterium or Bacillus species; Telavancin; Vibativ
MeSH Terms: conditions — Infections; Bacteremia; Sepsis; Staphylococcal Infections | interventions — telavancin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Telavancin (Experimental): 10 or 7.5 mg/kg intravenous daily
  Interventions: Drug: Telavancin

INTERVENTIONS:
Drug: Telavancin — 10 mg/kg by vein once daily for patients with a creatinine clearance of more than 50 ml/min, and a dose of 7.5 mg/kg once daily for patients with a creatinine clearance of 30-50 ml/min.
  Other Names: Vibativ

SUMMARY:
The goal of this clinical research study is to learn if Vibativ (telavancin) can help to control blood stream infections (BSIs). The safety of this treatment will also be studied.

Objectives:

Evaluate the clinical efficacy and safety of Telavancin given for treatment of gram positive bacteremia in cancer patients (including neutropenics).

DETAILED DESCRIPTION:
The Study Drug:

Telavancin is an antibiotic designed to treat a variety of bacterial infections that are difficult to treat.

Central Venous Catheter (CVC):

A CVC is a sterile flexible tube could have been placed into a large vein while you were under local anesthesia.

If you have a certain type of infection, your doctor may decided to remove or exchange your CVC. The decision to remove or exchange the CVC and timing of the placement of the new CVC will be decided by your primary doctor.

If you are to get a new CVC, your doctor will explain this procedure to you in more detail, and you will be required to sign a separate consent form.

Study Treatment:

If you are found to be eligible to take part in this study, you will receive telavancin by vein over a period of 60 minutes once daily for at least 7 days and for up to 6 weeks. How long you receive the study drug will depend on the type of bacterial infection that you have and if your doctor thinks you may have a complicated bacterial infection of the blood.

If the doctor thinks that you have a mixed infection (2 or more certain types of bacteria), you may also be given another type of antibiotic (such as aztreonam, cefepime, imipenem, meropenem, ciprofloxacin hydrochloride, bactrim, piperacillin/tazobactam and/or amoxicillin/clavulanate).

If the doctor thinks it is needed, you will have an echocardiogram to check your heart function. This test will only be performed if you have a specific type of infection (to make sure you do not have inflammation in the lining of the heart). You will be asked about medications you are taking.

If you are discharged from the hospital before completing the study drug, you will be able to take the drug as an outpatient. Your primary doctor may arrange for you to receive medication at M. D. Anderson.

Study Visits:

Once a week:

* Blood (about 1 tablespoon) will be drawn for routine tests. It may be drawn from the CVC, if the CVC is still in place.
* The CVC exit site will be checked at each visit until you have no more signs or symptoms of infection.
* You will be asked about any symptoms or illnesses that you may have had since your last visit.

Every other day, blood (about 1 tablespoon) will be drawn to check for the infection until it no longer shows signs of infection. Kidney function will be monitored by performing a blood test every 2 days for the first week and weekly after that.

Length of Study:

You can receive the study drug for up to 6 weeks. You will be taken off this study if the infection gets worse or any intolerable side effects occur.

End-of-Study Visit and Follow-up Visit:

You will need to return to MD Anderson for your end of treatment visit, within 7 days after you last dose of study drug. The end-of-study visit will occur within 7 days after your last dose of the study drug.

The follow-up visit will occur about 32 days (about 1 month) after your last dose of the study drug. At each of these visits, you will have the following exams/procedures performed.

* You will have a physical exam, including measurement of your vital signs.
* Blood (about 1 tablespoon) will be drawn for routine tests and to check for bacterial infection. The blood sample may be drawn from the CVC, if the CVC is still in place. The CVC exit site will be examined.
* You will be asked about any symptoms or illnesses that you may have had since your last visit.
* You will be asked about any drugs or therapies that you may be taking until the end of your treatment.
* If your infection recurs during the follow-up period, and if the doctor thinks it is needed, you will have an echocardiogram to check your heart function and to make sure you do not have inflammation in the lining of the heart.

This is an investigational study. Telavancin is FDA approved and commercially available for the treatment infections of the skin and soft tissue. Its use to treat blood infections in this study is investigational.

Up to 40 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with probable or definite diagnosis of uncomplicated gram positive bacteremia that have at least one positive blood culture including 20 patients with Staphylococcus aureus and the other 20 patients will include any of the following organism ( CNS, Enterococci, streptococci, pneumococci, Corynebacterium, and Propionibacterium or Bacillus species).If the positive blood culture involves a commensal skin organism such as CNS, Corynebacterium, Propionibacterium, Micrococcus and Bacillus, then at least > 100 colonies/ml will be required or a time to positivity =/< 16 hours (as it has been shown to reflect a high grade bacteremia), or two positive blood cultures. (Time to positivity of a blood culture bottle is recorded in the microbiology laboratory by the automatic culture detector (Bactec 9240 and Bactec Plus Aerobic/F; Becton Dickinson) which records culture positivity every 15 min according to changes in fluorescence related to microbial growth).
2. Patients must have at least two signs of sepsis from the list below, in any combination at any time, within 48 hours prior to Telavancin therapy: a. Core temperature =/>38.0 degrees C or =/<36.0 degrees C, measured orally, rectally, tympanic ally or via a central catheter. If auxiliary add 0.5 degrees C to the measured temperature; b. Pulse rate =/> 100 beats/min.; c. Respiratory rate =/> 20/min.; d. WBC count =/>12,000/mm^3, =/<4,000/mm or differential count showing >10% band forms; e. Systolic blood pressure =/<90 mm Hg. Patient will still be eligible for the study if the participants white blood cell count (WBC) is outside normal limits due to chemotherapy treatment or underlying conditions.
3. Male or non-pregnant, non-lactating females with an age of greater than or equal to 18 years.
4. Signed informed consent.
5. Female patients must be at no risk for pregnancy for one of the following reasons: - Postmenopausal for at least one year - Post-hysterectomy and/or post-bilateral ovariectomy - If of childbearing potential, having a negative serum human chorionic gonadotropin (hCG) pregnancy test with in 5 days prior to enrollment and be using a highly effective method of birth control throughout the course of the study. Reliable sexual abstinence throughout the course of the study is acceptable as a highly effective method of birth control for the purposes of this study.

Exclusion Criteria:

1. Estimated Serum Creatinine Clearance <30 mL/min (according to Cock-Gault-formula using ideal body weight) at the time gram positive bacteremia was diagnosed unless the patient is on dialysis.
2. Bilirubin >4x the upper limit of normal at the time gram positive bacteremia was diagnosed.
3. Treatment with an antibiotic, such as vancomycin, linezolid, tigecycline or Telavancin, effective against resistant gram positive bacterial infections, such as methicillin resistant staphylococci, for more than 48 hours within 72 hours of study medication initiation, unless treatment failed that is defined as a persistent fever and/or leukocytosis for 72 hours or longer of appropriate antibiotics treatment.
4. History of hypersensitivity to lipoglycopeptides.
5. Presence of deep-sited intravascular source of infection with same organism cultured from blood, e.g. endocarditis (as evidenced by vegetations on an echocardiogram), or septic thrombosis.
6. Presence of a prosthetic valve.
7. Oliguria defined as urine output of <20 cc/hour averaged over 24 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Issam Raad, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Chaftari AM, Hachem R, Jordan M, Garoge K, Al Hamal Z, El Zakhem A, Viola GM, Granwehr B, Mulanovich V, Gagel A, Reitzel R, Yousif A, Jiang Y, Raad I. Case-Control Study of Telavancin as an Alternative Treatment for Gram-Positive Bloodstream Infections in Patients with Cancer. Antimicrob Agents Chemother. 2015 Oct 19;60(1):239-44. doi: 10.1128/AAC.00617-15. Print 2016 Jan. PMID 26482312
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: March 2011 and May 2013. All recruitment done at The University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: One participant was excluded from the study because of a failed screening test result and did not receive treatment.
Groups:
- Telavancin: Telavancin 10 mg/kg intravenous (IV) once daily for patients with a creatinine clearance of more than 50 ml/min, and a dose of 7.5 mg/kg once daily for patients with a creatinine clearance of 30-50 ml/min.
Period: Overall Study
Arm/Group | Telavancin
Started | 39
Completed | 25
Not Completed | 14
Not completed — Lack of Efficacy | 5
Not completed — Adverse Event | 5
Not completed — Death | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Telavancin
Number analyzed (Participants) | 39
Age, Continuous [Median (Full Range); unit: years] | 61 [20 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 21
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Patient Clinical Response to Telavancin
Description: Clinical response assessed: Cure (No fever/chills or symptoms + eradication causing organism); Improvement (Resolution local/systemic symptoms + no new systemic antibacterial treatment); Failure (IF one or more following: Persistence 1+ symptoms [fever/chills] + new systemic anti gram positive treatment, > 72 hours after initiation study drug; or Relapse within 1 month completing antibiotic therapy; or Development of deep-seated infection not previously assessed); Indeterminate (clinical signs and symptoms cannot be assessed).
Time Frame: From baseline up to 6 weeks, assessed every 7 days
Population: Three patients received <72 hours of Telavancin treatment and therefore were excluded from the efficacy analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Telavancin
Number analyzed (Participants) | 36
Participants | 32

ADVERSE EVENTS:
Time Frame: Adverse event collected over duration of study drug therapy at least 7 days and up to 6 weeks.
Arm/Group | Telavancin
All-Cause Mortality (participants affected / at risk) | 7/39
Serious Adverse Events (participants affected / at risk) | 15/39
Other Adverse Events (participants affected / at risk) | 31/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Telavancin (N=39)
Intracerebellar bleed (Nervous system disorders) | 1
Fever (Infections and infestations) | 1
Neutropenic fever (Blood and lymphatic system disorders) | 3
Intraabdominal hemorrhage (Gastrointestinal disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Hypotension (Cardiac disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 4
Acute Renal Injury (Renal and urinary disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 1
Tumor lysis syndrome (Blood and lymphatic system disorders) | 1
Bowel obstruction (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Pneumonia (Infections and infestations) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Bloodstream infection (Infections and infestations) | 1
Acute coronary syndrome (Cardiac disorders) | 1
Neuropathy (Nervous system disorders) | 1
Sepsis (Infections and infestations) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telavancin (N=39)
Abdominal pain (General disorders) | 2 (2)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 1 (1)
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 10 (13)
Anorexia (Gastrointestinal disorders) | 2 (2)
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 1 (1)
Blood and lymphatic system disorders - (Other) (Blood and lymphatic system disorders) | 2 (2)
Blood bilirubin increased (Investigations) | 2 (2)
Bruising (Blood and lymphatic system disorders) | 1 (1)
Confusion (Nervous system disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Creatinine increased (Investigations) | 8 (10)
Diarrhea (Gastrointestinal disorders) | 5 (5)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Edema face (Skin and subcutaneous tissue disorders) | 1 (1)
Edema limbs (Musculoskeletal and connective tissue disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Esophageal pain (Gastrointestinal disorders) | 1 (1)
Eye disorders - (Other) (Eye disorders) | 2 (2) — Inflammed
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5)
Fever (Investigations) | 5 (7)
Floaters (Eye disorders) | 1 (1)
Gastrointestinal disorders (Gastrointestinal disorders) | 3 (4)
Hematoma (Vascular disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Hepatic hemorrhage (Hepatobiliary disorders) | 1 (1)
Hepatitis viral (Infections and infestations) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 7 (8)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (4)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (5)
Hypotension (Vascular disorders) | 1 (1)
Infections and infestations - (Other) (Infections and infestations) | 2 (2)
Intracranial hemorrhage (Nervous system disorders) | 1 (2)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 5 (5)
Neutrophil count decreased (Investigations) | 6 (9)
Pelvic infection (Infections and infestations) | 1 (1)
Platelet count decreased (Investigations) | 9 (15)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Psychiatric disorders - (Other) (Psychiatric disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Scrotal infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1)
Skin and subcutaneous tissue disorders - (Other) (Skin and subcutaneous tissue disorders) | 1 (1)
Skin infection (Skin and subcutaneous tissue disorders) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Surgical and medical procedures - (Other) (Surgical and medical procedures) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1)
Vascular access complication (Vascular disorders) | 1 (1)
White blood cell decreased (Investigations) | 8 (11)
Wound infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes